CLINICAL TRIAL: NCT00002024
Title: Ganciclovir: Compassionate Use in Patients With Serious or Life-Threatening Cytomegalovirus Infections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 029B; ICM 1257A
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1989-09

CONDITIONS: Cytomegalovirus Infections; HIV Infections
Keywords: AIDS-Related Opportunistic Infections; Immune Tolerance; Ganciclovir; Drugs, Investigational; Cytomegalovirus Infections; Acquired Immunodeficiency Syndrome
MeSH Terms: conditions — Cytomegalovirus Infections; HIV Infections; AIDS-Related Opportunistic Infections; Multiple Acyl Coenzyme A Dehydrogenase Deficiency; Acquired Immunodeficiency Syndrome | interventions — Ganciclovir

INTERVENTIONS:
Drug: Ganciclovir

SUMMARY:
To provide ganciclovir on a compassionate use basis to immunocompromised patients with serious cytomegalovirus (CMV) infections and to study safety and efficacy in this patient population.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Topical acyclovir.

Exclusion Criteria

Co-existing Condition:

Patients with the following are excluded:

* Mild to moderate cytomegalovirus (CMV) infections that fail to satisfy the clinical severity criteria.
* Transplant where a trial reduction of immunosuppressive drug treatment is not feasible.
* Congenital or neonatal CMV infections where there is not documented congenital or acquired immunodeficiency.
* Neutropenia unless it is pre-existing.
* Thrombocytopenia unless it is pre-existing.

Concurrent Medication:

Excluded:

* Other myelosuppressive drugs such as cancer chemotherapy agents, interferon, foscarnet, or nucleoside analogs.

Patients with the following are excluded:

* Mild to moderate cytomegalovirus (CMV) infections that fail to satisfy the clinical severity criteria.
* Transplant where a trial reduction of immunosuppressive drug treatment is not feasible.
* Congenital or neonatal CMV infections where there is not documented congenital or acquired immunodeficiency.
* Neutropenia unless it is pre-existing.
* Thrombocytopenia unless it is pre-existing.

Patients must be immunocompromised with a serious cytomegalovirus (CMV) infection. This would include pneumonia, gastrointestinal disease, hepatitis, or other organ-specific disease or severe wasting syndrome. Patients with pre-existing neutropenia or thrombocytopenia, and immediate life-threatening disease can be included if the investigator believes that delay in starting ganciclovir therapy is not advisable. In such patients, the investigator must advise the patient of the risk of further marrow suppression and the increased risk of infection or bleeding; and the patient must sign an amended informed consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Roche Global Development - Palo Alto, Palo Alto, California, United States

REFERENCES:
- [Background] Spector SA, McKinley GF, Lalezari JP, Samo T, Andruczk R, Follansbee S, Sparti PD, Havlir DV, Simpson G, Buhles W, Wong R, Stempien M. Oral ganciclovir for the prevention of cytomegalovirus disease in persons with AIDS. Roche Cooperative Oral Ganciclovir Study Group. N Engl J Med. 1996 Jun 6;334(23):1491-7. doi: 10.1056/NEJM199606063342302. PMID 8618603